CLINICAL TRIAL: NCT06194292
Title: Work in Green Spaces and Musculoskeletal Disorders: a Cross-sectional Descriptive Study Within the Territorial Civil Service of the Grand Est (France)
Brief Title: Work in Green Spaces and Musculoskeletal Disorders
Acronym: TEVTMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8959
Record Dates: First submitted 2023-12-15; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Musculoskeletal Disorders
Keywords: Musculoskeletal disorders; Osteoarticular
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Musculoskeletal disorders (MSDs) of the limbs and spine are painful conditions of the periarticular soft tissues (muscles, tendons, vessels, etc.) and peripheral nerves secondary to overuse of occupational origin.

They can manifest as pain (the most common symptom), discomfort, stiffness, loss of precision in movements or loss of strength. The lumbar spine and upper limbs are the parts of the body most frequently affected by MSDs.

MSDs have a multifactorial origin that can be separated into 2 categories: factors linked to the individual (age, sex, medical history) and factors linked to the work environment (biomechanical constraints, work organization, psychosocial risks).

MSDs are the leading cause of compensated occupational illnesses in France (86% of occupational illnesses in 2021, according to the Health Insurance annual report), particularly in the agricultural sector to which the majority of professions in green spaces belong. . If, in the Grand Est of France, the prevalence of employees exposed to physical risks decreased in the majority of sectors of activity between 1994 and 2017, we note at the same time a slight increase in the prevalence in the agricultural sector over this period. same period (6% in 2017 compared to 3.7% in 1994, SUMER 2017 survey).

Concerning the current context in France, the green spaces sector has undergone changes in recent years following the national implementation of the Ecophyto plan in 2008 (updated in 2015 then in 2018). This plan, the latest version of which is called Ecophyto 2+, aims to reduce the use of plant protection products by 50% by 2025. At the same time, the use of plant protection products for the maintenance of green spaces, forests, roads and walks have been prohibited by the Labbé law since January 1, 2017. In this context, and given the absence of recent data from the literature on this subject in France, the investigator wishes to carry out an inventory recent physical and organizational constraints, as well as the prevalence of MSDs, in the green space sector (targeting more particularly in its study the green spaces of the Territorial Civil Service of the Grand Est)

ELIGIBILITY:
Inclusion Criteria:

* Major subject from 18 to 62 years old
* Subject working in the service of green spaces in the Territorial Civil Service in a city in the Grand Est, active when the study was carried out
* Subject agreeing to participate in the study
* Subject with sufficient command of the French language to understand the self-questionnaire

Exclusion Criteria:

* Subject not wishing to participate in the study
* Subject on sick leave
* Subject under 18 years old or over 62 years old
* Subject under guardianship or curatorship
* Subject under judicial protection

Ages: 18 Years to 62 Years | Sex: All
Age Groups: Adult
Study Population: Major subject from 18 to 62 years old working in the service of green spaces in the Territorial Civil Service in a city in the Grand Est, active when the study was carried out
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the working conditions of green space maintenance workers leading to musculoskeletal disorders | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle - Médecine de Travail - CHU de Strasbourg - France, Strasbourg, France